CLINICAL TRIAL: NCT01074528
Title: Mindfulness Based Stress Reduction: Supportive Treatment for Adult Patients With Cancer and Their Partners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Belgian Federal Public Service, Food Chain Safety and Environment (Other Government)
Responsible Party: Principal Investigator, Prof. Dr. Christiaan Schotte, Professor, Belgian Federal Public Service, Food Chain Safety and Environment
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SCV2010
Record Dates: First submitted 2010-02-18; First posted 2010-02-24 (Estimated); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Cancer
Keywords: cancer patients; relatives or partners of cancer patients
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- mindfulness based stress reduction (Experimental): 8-week mindfulness based stress reduction program
  Interventions: Behavioral: mindfulness based stress reduction program
- control group (No Intervention): patients who have to wait before entering the MBSR program or who do not want to follow this program

INTERVENTIONS:
Behavioral: mindfulness based stress reduction program — 8-week mindfulness training program
  Other Names: MBSR
  Arms: mindfulness based stress reduction

SUMMARY:
The main purpose of this study is to evaluate the effects of the Mindfulness Based Stress Reduction (MBSR) training program that is offered in the investigator hospital, more specifically on quality of life, coping strategies and partner relationship by using questionnaires. To asses the possible impact of this treatment on the latter domain, partners of the patients with a cancer diagnosis are invited to join the training program.

DETAILED DESCRIPTION:
Patients with breast cancer often experience anxiety, depression, stress and reduced quality of life. As such, there is an increased interest in the implementation of the Mindfulness-Based Stress Reduction program as an additional supportive treatment. MBSR is a structured group program that aims at reducing stress levels by enhancing awareness of the present moment in combination with a non-judgemental attitude.

The study evaluates the effects of an 8-week MBSR program on quality of life, mood, depression, stress and coping skills in breast cancer patients.

Breast cancer patients of the Breast Clinic of the Universitair Ziekenhuis Brussel participate in the MBSR program. Before and after the training program patients filled out questionnaires evaluating quality of life, coping skills, emotional functioning, stress and aspects of mindfulness.

ELIGIBILITY:
Inclusion Criteria:

For patients:

* Cancer diagnosis
* Between the age of 18 until 70
* Dutch speaking

For partners:

* between the age of 18 until 70
* dutch speaking

Exclusion Criteria:

for patients and partners:

* Ongoing radiation therapy
* Psychiatric disorders
* Previous experience with mindfulness or meditation related techniques
* Pregnancy
* No or insufficient understanding of the Dutch language

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2010-04; Primary Completion 2017-04 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
quality of life (FACT) before training | day 1
Quality of life (FACT) after training | day 48

SECONDARY OUTCOMES:
Cancer Coping Questionnaire (CCQ) | day 1
Profile Of Mood Scale (POMS) | day 1
Perceived Stress Scale (PSS) | day 1
Freiburg Mindfulness Scale | day 1
Cancer Coping Questionnaire (CCQ) | day 48
Profile of Mood Scale (POMS) | day 48
Perceived Stress Scale (PSS) | day 48
Freiburg Mindfulness Inventory (FMI) | day48

CONTACTS AND LOCATIONS:
Overall Officials: Christiaan Schotte, PhD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- UZ Brussel, Brussels, Belgium